CLINICAL TRIAL: NCT05491694
Title: To Evaluate the Efficacy and Safety of Toripalimab Combined With Chemotherapy (Epirubicin + Cyclophosphamide → Nab-paclitaxel + Carboplatin) in the Neoadjuvant Treatment of Triple-negative Breast Cancer After High-intensity Focused Ultrasound (HIFU) Induction
Brief Title: To Evaluate the Efficacy of Toripalimab Combined With Chemotherapy After HIFU Induction in the Treatment of Early Triple-negative Breast Cancer
Acronym: HIFU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shui Wang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU202207
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — toripalimab; Epirubicin; Cyclophosphamide; Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU+Toripalimab+Chemotherapy (Experimental): High Intensity Focused Ultrasoun， followed by Toripalimab 240 mg + epirubicin 90 mg/m2 + cyclophosphamide 600 mg/m2 × 4 cycles → Toripalimab240 mg + carboplatin AUC 5 + nab-paclitaxel 260 mg/m2 IVD × 4 cycles every 3 weeks for 8 doses.
  Interventions: Drug: Toripalimab; Drug: Epirubicin; Procedure: High Intensity Focused Ultrasoun; Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg
Drug: Epirubicin — 90mg/m2，IVD，q3w
Procedure: High Intensity Focused Ultrasoun — HIFU treatment at lesion site
Drug: Cyclophosphamide — 600mg/m2，IVD，q3w
Drug: Carboplatin — AUC 5，IVD，q3w
Drug: Nab-paclitaxel — 260mg/m2，IVD，q3w

SUMMARY:
To investigate the efficacy and safety of terbinumab combined with chemotherapy (epirubicin + cyclophosphamide → nab-paclitaxel + carboplatin) in neoadjuvant therapy of triple-negative breast cancer after HIFU.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 years who require a negative pregnancy test for premenopausal and perimenopausal patients and promise to take reliable contraceptive measures during treatment;
2. Histopathologically confirmed breast cancer patients who are negative for estrogen receptor (ER), progesterone receptor (PR), and HER-2 by immunohistochemistry; positive PD-L1 expression in tumor cells (≥ 1%);
3. triple-negative breast cancer patients without distant metastasis;
4. According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, they have at least one evaluable target lesion;
5. ECOG PS score: 0 - 1;
6. New York Heart Association (NYHA) functional class I;
7. Electrocardiogram without myocardial ischemia, echocardiography LVEF > 55%, cardiac markers: cardiac troponin I (cTnI) and brain natriuretic peptide (BNP) test values within the normal range;
8. Normal major organ function, Meet the following criteria:

WBC ≥ 4.0 × 10 9/L,Neutrophil count (ANC) ≥ 1.5 × 10 9/L; platelet ≥ 100 × 10 9/L; hemoglobin ≥ 10 g/dL; serum creatinine ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) ≤ 2.5 × ULN; alanine aminotransferase (ALT) ≤ 2.5 × ULN; total bilirubin ≤ 1.5 × ULN; serum creatinine ≤ 1.5 × ULN;

9) The subject is able to understand the study procedures, voluntarily join the study, sign the informed consent form, have good compliance, and cooperate with the follow-up.

-

Exclusion Criteria:

1. Patients during pregnancy and lactation, women of childbearing age who refuse to take effective contraceptive measures during the study period; Patients with peripheral nervous system disorders caused by diseases or those with a history of significant mental disorders and central nervous system disorders;
2. Serious or uncontrolled infections that may affect the evaluation of study treatment or study results, including but not limited to: active hepatitis virus infection, human immunodeficiency virus (HIV) antibody positive, lung infection, etc.;
3. Known allergy to the active ingredients or other components of the study drug or surgical contraindications;
4. In addition to cured basal cell carcinoma of the skin and cured cervical carcinoma in situ, other cancers are disease-free for less than 5 years;
5. Severe liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, active gastrointestinal ulcers and other need treatment;
6. Need to receive other anti-tumor therapy (except ovarian function inhibitors) during neoadjuvant therapy as judged by the investigator;
7. Patients who are participating in other clinical trials within one month;
8. Patients with severe heart disease or discomfort, Expected intolerance to chemotherapy,Including, but not limited to: a. fatal arrhythmia or higher grade atrioventricular block (second-degree type 2 [Mobitz 2] atrioventricular block or third-degree atrioventricular block); b. unstable angina pectoris; c. clinically significant valvular heart disease; d. transmural myocardial infarction on electrocardiogram; e. uncontrolled hypertension;
9. any other condition that in the opinion of the investigator would make the patient inappropriate for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pCR | 6 months
  Pathologic complete response rate